CLINICAL TRIAL: NCT00382226
Title: IOP-Lowering Efficacy of Brinzolamide 1.0% Added to Travoprost 0.004%/Timolol 0.5% Fixed Combination as Adjunctive Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM-05-10
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2008-04

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — brinzolamide

INTERVENTIONS:
Drug: Azopt

SUMMARY:
Uncontrolled glaucoma patients being treated with a prostaglandin agent alone or in combination with adjunctive drugs in fixed or unfixed combinations, will be switched from their current therapy to travoprost/timolol fixed combination and either Azopt or placebo

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma

Exclusion Criteria:

* Under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
IOP lowering

SECONDARY OUTCOMES:
safety

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jasek, Study Director — Alcon Research
Locations (1):
- Sydney Study Site, Sydney, New South Wales, Australia

REFERENCES:
- [Result] Goldberg I, Crowston JG, Jasek MC, Stewart JA, Stewart WC; ADAPT Study Investigator Group. Intraocular pressure-lowering efficacy of brinzolamide when added to travoprost/timolol fixed combination as adjunctive therapy. J Glaucoma. 2012 Jan;21(1):55-9. doi: 10.1097/IJG.0b013e3181fc8142. PMID 21048504